CLINICAL TRIAL: NCT05706987
Title: Does Lidocaine Reduce Patient Moving Which Affect the Procedure Proceeding and Improves Surgeon Satisfaction in Labiaplasty
Brief Title: Lidocaine Improves Satisfaction in Labiaplasty
Acronym: anesthetics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20220178
Record Dates: First submitted 2022-11-30; First posted 2023-01-31 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2022-11

CONDITIONS: Lidocaine
Keywords: Lidocaine; labiaplasty
MeSH Terms: interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine infusion (Experimental): intravenous lidocaine infusion 1.5mg/kg/hr (ideal body weight) during labiaplasty
  Interventions: Drug: Lidocaine
- normal saline infusion (Placebo Comparator): equal volume of normal saline infusion during labiaplasty
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine — continuous lidocaine infusion perioperatively
  Arms: lidocaine infusion
Drug: Normal saline — normal saline
  Arms: normal saline infusion

SUMMARY:
1.Written informed consent must be obtained before any study specific procedures are undertaken.Qualified participants were identified at the pre-anesthesia evaluation clinic or ward.

2.80 patients with American Society of Anesthesiologists (ASA) score of I-II in our medical center scheduled to undergo elective surgery for hypertrophy of labia minor with MAC. Patients were randomized 1:1 into the Group 1 (normal saline) or Group 2 (lidocaine 1.5 mg/kg/hr, ideal body weight) by using a table of random, computer-generated digits in sealed and numbered envelopes by an anesthesiologist. All surgical procedure was performed by the same surgeon and the anesthetic data was recorded by a nurse anesthetist. All patients were fasted overnight before the procedure, and no medications were allowed before induction of anesthesia. Standard monitoring, such as non-invasive arterial blood pressure, electrocardiography (lead II), pulse oximetry, end-tidal carbon dioxide pressure (EtCO2) was applied for each patient. Participants were pre-oxygenated and adequately maintained with 100% oxygen at 3 L/min via a nasal cannula during the entire procedure. During anesthesia induction, all patients received intravenous fentanyl 0.5-1 mcg/kg, continuous infusion of propofol with target-controlled infusion (TCI; Fresenius Orchestra Primea; Fresenius Kabi AG, Bad Homburg, Germany) with the Ce of 4.0 mcg/mL and parecoxib. In addition, continuous infusion of equal volume normal saline and lidocaine 1.5 mg/kg/hr (ideal body weight) in group I and 2, respectively. In all patients, maintenance of the Ce of propofol was adjusted upward or downward by 0.5 mcg/mL to keep patient adequate sedation with acceptable pain (remaining moveless). If upward 2 times of propofol and the patient still move which affect the surgical procedure, fentanyl 0.5 mcg/kg was prescribed, and mean arterial pressure (MAP) and heart rate (HR) within baseline levels. As soon as the last suture, the propofol and lidocaine were discontinued. After the procedure, all patients were sent to the PACU for further care under clear consciousness.

DETAILED DESCRIPTION:
Patients were monitored for MBP, HR, peripheral oxygen saturation (SpO2), respiratory rate (RR), EtCO2, Ce of propofol, BIS values, OAA/S at the T1: before anesthesia induction, T2: time of the skin incision, T3: 15 minutes after the skin incision, T4: 30 minutes after the skin incision, T5: 45 minutes after the skin incision, T6: time of the beginning skin suture, and T7: time of the end of procedure. Collected data also include the time that the surgery ended, the total usage of propofol and fentanyl, the frequency to adjustment of TCI, times of patient move affect the procedure, and the surgeon's satisfaction. At PACU, patients were monitored for HR, MBP, SpO2, RR, NRS, RASS, length of stay, PONV and patient satisfaction (scoring 1-5).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-80 years old
2. ASA score I-II
3. receiving labiaplasty

Exclusion Criteria:

1. age < 20 years or older than 80 years
2. ASA score more than II
3. height <152 and >213 cm
4. body mass index > 35 kg/m2
5. allergy to midazolam and lidocaine
6. chronic use of opioid drugs

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
the alteration of total usage of propofol and fentanyl | about 1 hour (perioperatively)
  Comparing the treatment group with the control group the total infusion dose of propofol sedation and bolus intravenous fentanyl use perioperatively

SECONDARY OUTCOMES:
the alterations of total adverse events | up to 1 hour
  Comparing the total adverse events caused by propofol sedation or fentanyl analgesics such as apnea or hypoxemia between the treatment and the control group
postoperative patient's satisfaction after anesthesia | 1 hour after the surgery.
  Comparing the patient's satisfaction after anesthesia between the treatment group and the control group. The patient would be asked to score her satisfaction from 1-5, 1 as very dissatisfied, 2 as dissatisfied, 3 as neutral, 4 as satisfied and 5 as very satisfied.
the surgeon's satisfaction after anesthesia service | immediately after the surgery
  Comparing the surgeon's satisfaction after anesthesia service between the treatment group and the control group. The surgeon's satisfaction after anesthesia service would be calculated by scoring 1-5, 1 as very dissatisfied, 2 as dissatisfied, 3 as neutral, 4 as satisfied and 5 as very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Fu Wu, MD, Study Director — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan